CLINICAL TRIAL: NCT05053581
Title: Evaluation of Self-efficacy as a Predictor for CPAP-compliance in a OSAS-patients French Cohort
Acronym: SAFES
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Air Liquide Santé International (Industry)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2020/45
Record Dates: First submitted 2021-08-31; First posted 2021-09-22 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Sleep Apnea, Obstructive
Keywords: Continuous positive airway pressure therapy; Sleep Apnea; Obstructive Sleep Apnea Syndrome
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — Patients will complete 7 questionnaires at inclusion (T0) and 1,3 and 6 months after start of CPAP treatment

SUMMARY:
Continuous positive airway pressure (CPAP) is the reference treatment for obstructive sleep apnea syndrome (OSAS) and is effective in improving symptoms of OSAS, reducing risk of accidents and improving quality of life. However, CPAP use is less than optimal. Recommended use is between 6-8 hour per night and a common clinical and empiric benchmark has been defined for CPAP use as an average of 4h per night for 70% of the night. Approximatively 30% of patients discontinue CPAP treatment during the first weeks. Thus, it is very important to identify the factors that influence CPAP adherence during the first weeks of treatment.

Biomedical factors, in particular nose respiratory abnormalities, somnolence complaints and insomnia complaints, have been widely studied but explain only 4 to 25 % of the variance in CPAP use. Interestingly, "self-efficacy" (the confidence to engage in a treatment), was found to explain more than 30 % of the variance in CPAP use.

The SEMSA (Self Efficacy in Sleep apnea) questionnaire is the instrument to investigate self-efficacy related to OSAS and CPAP that has received the most attention. Retrospective studies showed that the factor "self-efficacy" of the SEMSA was related to poor CPAP adherence. Prospective studies showed that the factor "self-efficacy" of the SEMSA at baseline was associated with future CPAP use when it was completed after education information.

A French version of the SEMSA has been validated by investigators in a retrospective study. They have confirmed in France that the factor "self-efficacy" of the SEMSA was related to poor CPAP adherence. No prospective study using the SEMSA has been conducted in French patients with OSAS treated with CPAP. Given the specificity of the French health care system and home care system, it is thus important to evaluate the predictive value of self-efficacy on CPAP adherence in France. The generation of predictive model would enable pretreatment prediction of those likely to have difficulty with CPAP adherence, and would serve as the basis for the development of maximally effective interventions in order to enhance CPAP adherence by patients with OSAS.

DETAILED DESCRIPTION:
Using a prospective design, investigators aim to examine the following factors: pre-treatment demographic factors, sleep clinical factors (Somnolence complaints with ESS questionnaire and Insomnia complaints with ISI questionnaire), patients' perceptions of self-efficacy (SEMSA questionnaire), and nose respiratory complaints (NOSE questionnaire).

The objective is to investigate if self-efficacy would be the best predictor of CPAP use during the first month of treatment and at 3 and 6 months after treatment beginning. Impact of demographic factors, sleep and nose complaints will be taken into account.

The study intend to recruit at the sleep clinic 150 patients with newly diagnosed Obstructive Sleep Apnea Syndrome for whom CPAP treatment is indicated.

During the consultation of CPAP treatment initiation, the investigator will present the study and give the informed notice. If the patient agrees to participate, the investigator will notify the non-opposition of the patient in the medical file and confirm eligibility criteria. The patient will then complete 4 questionnaires (ISI, ESS, SEMSA, NOSE).

After initiation of CPAP treatment, the same questionnaires will be sent to the patient 1 month, 3 and 6 months after treatment beginning.

A Clinical Research Associate will call the patient to ensure the completion of questionnaires or in case of missing or incomplete data.

The result of this study will give the opportunity to have a predictive model that enable pretreatment prediction of those likely to have difficulty with CPAP use, and would serve as the basis for the development of maximally effective interventions in order to enhance CPAP adherence by patients with OSAS.

ELIGIBILITY:
Inclusion Criteria:

* Patients with new OSAS-diagnosed (Apnea-Hypopnea Index≥ 15) with CPAP as intended treatment
* Patients agreeing follow-up by telemonitoring
* Age between 18 and 65 years
* Affiliated person or beneficiary of a social security scheme
* Informed and expressed his/her non-opposition to engage in the study

Exclusion Criteria:

* Night-workers or shift-workers
* Current psychiatric disorder (mood disorders, anxiety disorders, psychosis, dependence interfering with nocturnal sleep) assessed by the investigator during medical interview
* Current neurologic disorders interfering with sleep (for example: neurodegeneratives diseases, stroke, epilepsy) assessed by the investigator during medical interview
* Uncontrolled cardiovascular or respiratory disorders
* Pregnant women or breastfeeding mother.
* Person under guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with new OSAS-diagnosed with CPAP as intended treatment
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2022-05-18 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
CPAP Compliance M1 | Month 1 after CPAP initiation (inclusion)
  Mean of the number of daily hours using CPAP on 30 days of data collection by telemonitoring before administration of M1 follow-up questionnaire

SECONDARY OUTCOMES:
CPAP Compliance M3 and M6 | Month 3 and Month 6 after CPAP initiation (inclusion)
  Mean of the number of daily hours using CPAP on 30 days of data collection by telemonitoring
OSAS consequences et risk perception | CPAP initiation (inclusion), then Month 1, Month 3, and Month 6 after CPAP initiation
  Factor "perception of the consequences and risks of OSAS" of SEMSA questionnaire
Expected benefits of CPAP | CPAP initiation (inclusion), then Month 1, Month 3, and Month 6 after CPAP initiation
  Factor "perception of the expected benefits of CPAP" of SEMSA questionnaire.
Demographics before treatment | CPAP initiation (inclusion)
  Demographic factors before CPAP treatment: age, sex, socio-professional category, marital status, body mass index, cardiovascular disorders, metabolic disorders, antidepressant treatments
Insomnia Severity Index (ISI) | CPAP initiation (inclusion), then Month 1, Month 3, and Month 6 after CPAP initiation
  Insomnia complaints with ISI questionnaire
Epworth Sleepiness Scale (ESS) score | CPAP initiation (inclusion), then Month 1, Month 3, and Month 6 after CPAP initiation
  Sleepiness complaints with ESS (Epworth Sleepiness Scale) questionnaire. The ESS score can range from 0 to 24. The higher the ESS score, the higher that person's average sleep propensity in daily life, or their 'daytime sleepiness'.
Hypersomnia Severity Index (HSI) | CPAP initiation (inclusion), then Month 1, Month 3, and Month 6 after CPAP initiation
  Sleepiness complaints with HSI questionnaire
Nasal Respiratory complaints | CPAP initiation (inclusion), then Month 1, Month 3, and Month 6 after CPAP initiation
  Nasal Respiratory complaints measured by NOSE questionnaire
Depression symptoms | CPAP initiation (inclusion), then Month 1, Month 3, and Month 6 after CPAP initiation
  Depression symptoms measured by PHQ-4 questionnaire
Anxiety symptoms | CPAP initiation (inclusion), then Month 1, Month 3, and Month 6 after CPAP initiation
  Anxiety symptoms measured by PHQ-4 questionnaire
Reasons for CPAP initiation | CPAP initiation (inclusion)
  Factors which led up to CPAP initiation

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Bordeaux, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No